CLINICAL TRIAL: NCT05426993
Title: Investigation of the Effects of Metabolic Syndrome on the Results of Complex Decongestive Physiotherapy in Lymphedema Patients
Brief Title: Effect of Metabolic Syndrome on Complex Decongestive Physiotherapy Outcomes in Lymphedema Patients
Status: Completed | Type: Observational
Sponsor: Gulhane School of Medicine (Other)
Responsible Party: Principal Investigator, Mustafa Ertuğrul Yaşa, Assocc. Prof., Gulhane School of Medicine
Other Study IDs: E2-22-1805
Record Dates: First submitted 2022-06-16; First posted 2022-06-22 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-12

CONDITIONS: Lymphedema
Keywords: lymphedema; metabolic syndrome
MeSH Terms: conditions — Lymphedema; Metabolic Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients diagnosed with lymphedema with metabolic syndrome: Demographic information of the patients (age, height, weight, occupation, history), comorbid diseases (hypertension, diabetes, cardiac problems, circulatory problems, thyroid dysfunction), operation date, operation type, affected extremity, type of lymphedema will be recorded. In addition to these, mental status, edema and quality of life assessments will also be made.
  As a treatment, extremity volume and quality of life evaluations will be made before and after the first phase of CDT (manual lymphatic drainage, skin care, compression therapy and exercises) for 3 weeks.
  Interventions: Other: Complex decongestive physiotherapy
- Patients diagnosed with lymphedema without metabolic syndrome: Demographic information of the patients (age, height, weight, occupation, history), comorbid diseases (hypertension, diabetes, cardiac problems, circulatory problems, thyroid dysfunction), operation date, operation type, affected extremity, type of lymphedema will be recorded. In addition to these, mental status, edema and quality of life assessments will also be made.
  As a treatment, extremity volume and quality of life evaluations will be made before and after the first phase of CDT (manual lymphatic drainage, skin care, compression therapy and exercises) for 3 weeks.
  Interventions: Other: Complex decongestive physiotherapy

INTERVENTIONS:
Other: Complex decongestive physiotherapy — CDT is a treatment approach consisting of manual lymph drainage, skin care, compression bandage and exercises.

SUMMARY:
As a result of our research, investigators could not find any study investigating the effectiveness of complex decongestive physiotherapy (KBF) in lymphedema patients with metabolic syndrome. Therefore, our aim is to compare the effectiveness of KBF in patients with and without metabolic syndrome.

DETAILED DESCRIPTION:
This study was planned to investigate the effects of metabolic syndrome seen in patients with lymphedema on the results of complex decongestive physiotherapy. Lymphedema is a chronic disease characterized by the accumulation of protein-rich fluid in the interstitial space. Among all the treatment approaches known in the field, Complex Decongestive Physiotherapy (CDT) is accepted as the gold standard in the treatment of lymphedema. CDT is a treatment approach consisting of manual lymph drainage, skin care, compression bandage and exercises. In clinical studies conducted to date, the effectiveness of CDFT in the treatment of lower and upper extremity lymphedema has been clearly demonstrated.

Metabolic syndrome is a medical term that describes the combination of various cardiovascular risk factors such as insulin resistance, impaired glucose tolerance or diabetes mellitus, obesity, abdominal fat accumulation, dyslipidemia, hypertension, and coronary artery disease. Obesity, the cardinal component of the metabolic syndrome, is a well-known risk factor for lymphedema, and increased body mass index (BMI) is associated with the frequency and severity of lymphedema. Obesity often accompanies lymphedema due to the effect of lymphedema and the characteristics of patients with lymphedema.

Our aim in this study, which was planned in the light of these data, is to examine whether the presence of metabolic syndrome in patients with lymphedema changes the effectiveness of CDT.

ELIGIBILITY:
Inclusion Criteria:

* Those between the ages of 18-65,
* To be diagnosed with lymphedema in the lower or upper extremities
* Volunteering to participate in the study
* Getting >24 points from the Standardized Mini mental test

Exclusion Criteria:

* Having a score of <24 on the Standardized Mini Mental Test
* Finding any problem preventing communication

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: As a result of the power analysis made with the help of the preliminary study data using the G*Power 3.0.10 program; with 90% power, 5% margin of error and f=0.27 effect size, a total of at least 40 samples were found to be sufficient (metabolic syndrome group: 20; control group: 20).
  Patients diagnosed with lymphedema by a specialist in our clinic will be divided into 2 groups as those with metabolic syndrome and those without metabolic syndrome.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2022-07-15 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2023-03-15 (Actual)

PRIMARY OUTCOMES:
Limb volume | 15.09.2022
  Edema evaluation will be made for the lower extremity from the lateral malleolus to the groin at 4 cm intervals. For the upper extremity, it will be made from the styloid process of the ulna to the axilla at intervals of 4 cm. The extremity volume will be determined from the values obtained with the help of the Frustrum formula.

SECONDARY OUTCOMES:
Life quality | 15.12.2022
  Quality of life will be evaluated with the Lymphedema Quality of Life Scale used routinely. This assessment, which was validated by Borman et al., consists of 21 questions under the sub-titles of Function, Body Image, Symptom, and Emotion. Scoring between 1 and 4 is made for the first 20 questions. The total score for each area is calculated by adding all the scores and dividing by the total number of questions answered. High scores indicate lower quality of life. The last question about overall quality of life is scored from 0 to 10. Higher scores indicate better quality of life

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Sciences, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pirincci CS, Mete O, Yasa ME, Dalyan M. A comparative evaluation of the efficacy of complete decongestive therapy in the treatment of unilateral breast cancer-related lymphedema with and without metabolic syndrome. Support Care Cancer. 2024 Jun 29;32(7):473. doi: 10.1007/s00520-024-08676-z. PMID 38949715